CLINICAL TRIAL: NCT04270149
Title: A Phase I Study of Cancer Peptides Plus GM-CSF and Adjuvant Following Completion of Prescribed Systemic Therapy of Estrogen Receptor Positive Breast Cancer
Brief Title: Cancer Peptides Plus GM-CSF and Adjuvant in Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Lyerly (Other)
Responsible Party: Sponsor-Investigator, Herbert Lyerly, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00104868
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; estrogen receptor; peptide vaccine; immunotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ESR1 peptide vaccine (Experimental): 200 mcg ESR1 peptides plus 1ml Montanide and 100 mcg GM-CSF administered subcutaneously weeks 0, 1, 2, 4, 5, 6 for a total of 6 injections.
  Interventions: Biological: ESR1 peptide vaccine

INTERVENTIONS:
Biological: ESR1 peptide vaccine — ESR1 peptides plus Montanide and GM-CSF

SUMMARY:
This is a phase I study looking at the safety of cancer peptides combined with adjuvant and GM-CSF in subjects with estrogen receptor (ESR) positive breast cancer. The primary objective of the study is to determine the safety of of the peptide vaccine. The secondary objective is to evaluate the immune response to the vaccine. The peptides used in this vaccine are derived from the estrogen receptor and are combined with the adjuvant Montanide ISA and GM-CSF to enhance their immune response. A peptide vaccine of these peptides may improve outcomes of patients with endocrine resistant breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, resected, breast cancer with one of the following characteristics:

pT3 or greater T stage with any N stage and M0 pTxN+M0 (i.e., N1,2 or 3)

* HLA A0201+ and tumor is ER+
* Patients must have completed any standard chemotherapy recommended by their physician. There must be at least 4 weeks from their last dose of chemotherapy (or surgery if no chemotherapy was given) prior to the first dose of study vaccine. There should be no more than 5 years from the time of completion of any chemotherapy, surgery or HER2 targeted therapy. Ongoing endocrine therapies are permitted as long as they have been administered for at least 3 months prior to study enrollment.
* Age ≥ 18 years.
* Heme: WBC ≥ 3000/microliter, hemoglobin ≥ 9 g/dL, platelets ≥ 80,000/microliter.
* Adequate, renal and hepatic function with serum creatinine < 1.5 mg/dL, bilirubin < 1.5 mg/dL (except a bilirubin of <2.0 will be permitted for patents with Gilbert's syndrome), SGOT/SGPT < 2 x upper limit of normal.
* Ability to understand and provide signed informed consent that fulfills Institutional Review Board's guidelines.

Exclusion Criteria:

* Subjects with concurrent chemotherapy, radiation therapy, or immunotherapy are excluded. There must be at least 4 weeks between these prior therapy and study treatment. Subjects must have recovered from all acute toxicities from prior treatment. Peripheral neuropathy grade 1 due to prior therapy will be permitted.
* Subjects may not have history of distant metastases.
* Subjects with a history of autoimmune disease, such as but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. A positive ANA (anti-nuclear antibody) test without other evidence of autoimmune disease will not exclude a subject for this study. A prior history of autoimmune hypothyroidism will not exclude a subject.
* Subjects with serious intercurrent chronic or acute illness, such as cardiac disease, (NYHA class III or IV), hepatic disease, or other illness considered by the Principal Investigator as unwarranted high risk for investigational drug treatment.
* Subjects with a medical or psychological impediment to probable compliance with the
* Concurrent (or within the last 5 years) second malignancy other than non-melanoma skin cancer, cervical carcinoma in situ, controlled carcinoma in situ of the cervix, or controlled superficial bladder cancer.
* Presence of an active acute or chronic infection including: an urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology). Subjects with HIV are excluded based on immuno-suppression, which may render them unable to respond to the vaccine; subjects with chronic hepatitis are excluded because of concern that hepatitis could be exacerbated by the injections.
* Subjects on steroid therapy (or other immuno-suppressives, such as azathioprine or cyclosporin A) are excluded on the basis of potential immune suppression. Subjects must have had 6 weeks of discontinuation of any steroid therapy (except that used as pre-medication for chemotherapy or contrast-enhanced studies) prior to enrollment.
* Subjects with allergies to any component of the vaccine
* Pregnant or nursing mothers.
* Subjects with acute or chronic skin disorders that will interfere with peptide injection into the skin of the extremities or subsequent assessment of potential skin reactions will be excluded.
* Splenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 44 days
  Safety

SECONDARY OUTCOMES:
detection of ESR mutant-specific memory T cells against at least one of the 5 immunizing peptides by Cytof analysis | 2 years
  Detection of memory T cells

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No